CLINICAL TRIAL: NCT06356493
Title: Prophylactic Occlusion Balloons of Both Internal Iliac Arteries in Caesarean Hysterectomy for Placenta Accreta Spectrum Disorder Reduces Blood Loss: a Retrospective Comparative Study
Brief Title: Prophylactic Occlusion Balloons of Both Internal Iliac Arteries in Caesarean Hysterectomy for PASD
Status: Completed | Type: Observational
Sponsor: Tunis University (Other)
Responsible Party: Principal Investigator, Haithem Aloui, university hospital assistant, Tunis University
Other Study IDs: OBIIA CMNT
Record Dates: First submitted 2024-03-30; First posted 2024-04-10 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Hemorrhage; Placenta Accreta Spectrum; Cesarean Section Complications
Keywords: haemorrhage; Placenta accreta spectrum disorder; caesarean hysterectomy; occlusion balloons; internal iliac artery
MeSH Terms: conditions — Hemorrhage; Placenta Accreta

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group1: Patients treated by caesarean hysterectomy without prior placement of prophylactic occlusion balloons of both internal iliac arteries
  Interventions: Procedure: caesarean hysterectomy without prior placement of prophylactic occlusion balloons of both internal iliac arteries
- Group2:: Patients treated by caesarean hysterectomy with prior placement of prophylactic occlusion balloons of both internal iliac arteries
  Interventions: Procedure: caesarean hysterectomy with prior placement of prophylactic occlusion balloons of both internal iliac arteries

INTERVENTIONS:
Procedure: caesarean hysterectomy with prior placement of prophylactic occlusion balloons of both internal iliac arteries — Preoperative placement of prophylactic occlusion balloons of both internal iliac arteries (OBIIA) was performed at radiology department. Access to the internal iliac arteries was achieved by retrograde transcutaneous introduction of hydrophilic sheath kits of 8.5 mm under fluoroscopic guidance from both femoral arteries. Once in the lumens of the two internal iliac arteries, the radiologist inflated the balloons until blood flow ceased. The pressure at which occlusion of both internal iliac arteries was achieved was recorded for subsequent replication in the operating room. The radiologist secured the two kits to the skin and applied a compressive dressing. The patient was then directly transferred to the operating room.
  Groups: Group2:
Procedure: caesarean hysterectomy without prior placement of prophylactic occlusion balloons of both internal iliac arteries — Caesarean hysterectomy was performed through a midline infraumbilical incision. The bladder-uterine peritoneum was dissected, followed by a vertical fundal hysterotomy away from the placenta, and the baby was delivered This was followed by clamping the umbilical cord and closure of the hysterotomy while leaving the placenta in situ without any attempt at traction or delivery and without oxytocin administration.
  We proceeded with the remaining steps of hysterectomy.
  Groups: Group1

SUMMARY:
The placenta accreta spectrum is a heterogeneous disorder due to abnormal placental invasion into the uterine wall putting at risk the lives of the patients by causing a massive hemorrhage. Its incidence is increasing due to the rise of the cesarean section. The management of this spectrum is multidisciplinary but not yet codified. Hysterectomy-caesarean, though hemostatic surgery, remains the standard Gold. Several adjuvant treatments have emerged in recent years to minimize the risk of bleeding and morbidity of these disorders including the internal-iliac prophylactic occlusion balloons.

The aim of the study is to demonstrate the effect of prophylactic occlusion balloons in both uterine iliac arteries in the management of placental accreta spectrum disorders.

DETAILED DESCRIPTION:
Study population:

In the study, the population was divided into two groups:

Group1: Patients treated by caesarean hysterectomy without prior placement of prophylactic occlusion balloons of both internal iliac arteries.

Group2: Patients treated by caesarean hysterectomy with prior placement of prophylactic occlusion balloons of both internal iliac arteries.

Service Protocol:

All patients received dexamethasone for foetal lung maturation. Preoperative placement of prophylactic occlusion balloons of both internal iliac arteries (OBIIA) was performed at radiology department. Access to the internal iliac arteries was achieved by retrograde transcutaneous introduction of hydrophilic sheath kits of 8.5 mm under fluoroscopic guidance from both femoral arteries. Once in the lumens of the two internal iliac arteries, the radiologist inflated the balloons until blood flow ceased. The pressure at which occlusion of both internal iliac arteries was achieved was recorded for subsequent replication in the operating room. The radiologist secured the two kits to the skin and applied a compressive dressing. The patient was then directly transferred to the operating room.

General anaesthesia was preferred. Blood loss was estimated by weighing surgical sponges and drapes and quantifying aspirated blood.

Initially, a JJ stent was inserted for both groups to limit urinary tract injuries. Caesarean hysterectomy was performed through a midline infraumbilical incision. The bladder-uterine peritoneum was dissected, followed by a vertical fundal hysterotomy away from the placenta, and the foetus was delivered. Inflation of the occlusion balloons of both internal iliac arteries was performed simultaneously with extraction by the radiologist. This was followed by clamping the umbilical cord and closure of the hysterotomy while leaving the placenta in situ without any attempt at traction or delivery and without oxytocin administration.

the surgeon proceeded with the remaining steps of hysterectomy. The radiologist deflated the balloons at the end of the hysterectomy. The inflation of the OBIIA did not exceed 60 minutes. Haemostasis was verified, and an intraperitoneal drainage system was installed. A video was developed summarizing the procedure in Group 2.

ELIGIBILITY:
Inclusion Criteria:

* placenta accreta spectrum disorder (PASD) confirmed by histopathological examination.
* caesarean hysterectomy.

Exclusion Criteria:

* placenta accreta suspected in MRI fundings but disproved in in histopathological examination.
* conservative treatment of PASD

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: We collected 38 patients who were divided into two groups: Group 1 (n=22), Group 2 (n=16).
Sampling Method: Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2020-01-02 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
calculated blood loss | peroperatively
  The blood losses were calculated by weighing the surgical drapes and compresses and quantifying the aspirated bleeding
Transfusion peroperatively | First 24 hours]
  peroperatively
Duration of surgery | peroperatively
  MINUTES
Postoperative hospital stay | up to 40 days postpartum
  DAYS
Postoperative transfer to the intensive care unit | up to 40 days postpartum
  NUMBER

SECONDARY OUTCOMES:
Morbidity | time from surgery up to 30 days postoperative
  surgical site infection, bladder injury, need for surgical revision, and pulmonary embolism

CONTACTS AND LOCATIONS:
Overall Officials: Haithem Aloui, Doctor, Principal Investigator — Tunis University Manar
Locations (2):
- Tunisia (2):
  - Haithem Aloui, Manouba, Nabeul Governorate
  - Haithem Aloui, Tunis, Nabeul Governorate

IPD SHARING:
Plan to Share IPD: Undecided